CLINICAL TRIAL: NCT00415532
Title: A Randomized, Controlled, Open-label Study Evaluating the Efficacy and Tolerability of AMG 531 Versus Medical Standard of Care as Chronic Therapy for Non-splenectomized Subjects With Immune (Idiopathic) Thrombocytopenic Purpura
Brief Title: Romiplostim (AMG 531) Versus Medical Standard of Care for Immune (Idiopathic) Thrombocytopenic Purpura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060131
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Thrombocytopenia; Thrombocytopenia in Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenic Purpura
Keywords: splenectomy; platelet; AMG 531; thrombopoietin; blood disorder; bleeding disorder; immune thrombocytopenic purpura; idiopathic thrombocytopenic purpura; immune (idiopathic) thrombocytopenic purpura; TPO; thrombopoietic protein
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura, Thrombocytopenic; Jacobs syndrome; Hematologic Diseases; Hemostatic Disorders | interventions — Inosine Triphosphate; romiplostim

ARMS (2):
- Romiplostim (Experimental): Romiplostim administered by subcutaneous injection once weekly at a starting dose of 3 μg/kg, adjusted to a maximum dose of 10 μg/kg to maintain a platelet count between 50 and 200 x 10^9/L for up to 52 weeks.
  Interventions: Biological: Romiplostim
- Standard of Care (Other): Medical standard of care treatments were selected and prescribed by the investigator according to standard institutional practices or therapeutic guidelines and administered for up to 52 weeks.
  Interventions: Drug: Medical Standard of Care for ITP

INTERVENTIONS:
Drug: Medical Standard of Care for ITP
  Arms: Standard of Care
Biological: Romiplostim
  Other Names: AMG 531
  Arms: Romiplostim

SUMMARY:
This is a phase 3b, multi-center, randomized, Standard of Care (SOC)-controlled, open-label, 52-week treatment study to compare romiplostim to medical SOC for Idiopathic Thrombocytopenia Purpura (ITP), with a 6-month Safety Follow-up. Patients randomized to romiplostim must complete the taper or discontinuation of medical SOC for ITP as soon as medically feasible after the initiation of romiplostim. After the completion or discontinuation of the study treatment period, any participant who does not transfer in to another romiplostim study will complete a 6-month Safety Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject has a diagnosis of Idiopathic Thrombocytopenia Purpura (ITP) according to the American Society of Hematology (ASH) guidelines
* If subject is > 60 years of age, subject has a written bone marrow biopsy report confirming the diagnosis of ITP
* Subject has received at least 1 prior therapy for ITP
* Subject has a platelet count < 50,000 or their platelet count falls to < 50,000 during or after a clinically-indicated taper or discontinuation of current ITP therapy
* Before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

* Subject has had a splenectomy for any reason
* Subject has an active malignancy
* Subject has a history of cancer, other than basal cell carcinoma or cervical carcinoma in situ, with treatment or active disease within 5 years
* Subject has a known history of bone marrow stem cell disorder
* Subject has participated in any study evaluating polyethylene glycol-conjugated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), recombinant human thrombopoietin (rHuTPO), AMG 531, or a thrombopoietic protein
* Subject is receiving other investigational agents or procedures
* Subject is currently enrolled in, or has completed within the last 30 days, another investigational device or drug study
* Subject is pregnant or breast feeding
* Subject is not using adequate contraceptive precautions
* Subject has known sensitivity to any recombinant E. coli-derived product
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and does not have a legally acceptable representative
* Subject has any kind of disorder that compromises the ability of the subject to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2008-11-07 (Actual); Study Completion 2009-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Kuter DJ, Mathias SD, Rummel M, Mandanas R, Giagounidis AA, Wang X, Deuson RR. Health-related quality of life in nonsplenectomized immune thrombocytopenia patients receiving romiplostim or medical standard of care. Am J Hematol. 2012 May;87(5):558-61. doi: 10.1002/ajh.23163. Epub 2012 Mar 28. PMID 22460421
- [Background] Kuter DJ, Rummel M, Boccia R, Macik BG, Pabinger I, Selleslag D, Rodeghiero F, Chong BH, Wang X, Berger DP. Romiplostim or standard of care in patients with immune thrombocytopenia. N Engl J Med. 2010 Nov 11;363(20):1889-99. doi: 10.1056/NEJMoa1002625. PMID 21067381
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 20-Dec-2006 Last Subject Enrolled: 01-Nov-2007
Period: Treatment Period
Arm/Group | Standard of Care | Romiplostim
Started | 77 | 157
Received Treatment | 75 | 154
Switched to Romiplostim Group | 2 | 0
Completed | 60 | 142
Not Completed | 17 | 15
Not completed — Adverse Event | 2 | 3
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Other | 2 | 2
Not completed — Ineligibility determined | 1 | 1
Not completed — Noncompliance | 1 | 1
Not completed — Requirement for alternative therapy | 1 | 0
Period: Safety Follow Up Period
Arm/Group | Standard of Care | Romiplostim
Started | 43 (Participants who completed the treatment period were not required to participate in this follow-up) | 30 (Participants who completed the treatment period were not required to participate in this follow-up)
Completed | 34 | 18
Not Completed | 9 | 12
Not completed — Adverse Event | 1 | 3
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other | 1 | 4
Not completed — Ineligibility determined | 1 | 1
Not completed — Noncompliance | 1 | 0
Not completed — Requirement for alternative therapy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Romiplostim | Total
Number analyzed (Participants) | 77 | 157 | 234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (19.3) | 54.8 (18.8) | 54.7 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 85 | 131
  Male | 31 | 72 | 103
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 69 | 137 | 206
  Black or African American | 0 | 6 | 6
  Hispanic or Latino | 5 | 9 | 14
  Asian (Chinese, Bangladeshi, Indian, Pakistani) | 1 | 5 | 6
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Splenectomy During 52-Week Treatment Period
Description: Occurrence of a splenectomy. Participants who discontinued study during the treatment period prior to reporting a splenectomy were considered as having had a splenectomy.
Time Frame: 52 weeks
Population: The Full Analysis set includes all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Participants
  Had splenectomy | 28 | 14
  Did not have splenectomy | 49 | 143
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Significant level is set at 0.05; Odds Ratio (OR) = 0.172, 95% CI [0.084 to 0.352]

2. Primary Outcome: Number of Participants With Treatment Failure During 52-Week Treatment Period
Description: Treatment failure was defined by platelet counts ≤ 20 x 10^9/L for 4 consecutive weeks at the highest recommended dose and schedule, a major bleeding event, or change in therapy due to an intolerable side effect or bleeding symptom.
Time Frame: 52 weeks
Population: Full analysis set. Participants who discontinued study during treatment period prior to experiencing treatment failure were considered as having had treatment failure.
Measure: Number; unit: Participants
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Participants
  Had treatment failure | 23 | 18
  Did not have treatment failure | 54 | 139
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — Significant level is set at 0.05; Odds Ratio (OR) = 0.307, 95% CI [0.154 to 0.611]

3. Secondary Outcome: Time to Splenectomy
Description: Time to splenectomy in days calculated from date of randomization to date of splenectomy, or censored at date of end of treatment visit if no splenectomy was done during treatment period.
Time Frame: 52 weeks
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
days | NA [NA to NA] — Median and 95% confidence interval could not be estimated due to the low number of patients with splenectomy (15). | NA [NA to NA] — Median and 95% confidence interval could not be estimated due to the low number of patients with splenectomy (2).

4. Secondary Outcome: Percentage of Participants With Platelet Response
Description: Platelet response was defined as platelet counts > 50 x 10^9/L, measured at each study visit (excluding those within 8 weeks of prior rescue medication use) up to the time of splenectomy or the end of initial treatment period, whichever occurred first.
Time Frame: Weeks 1-8, and Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Full analysis set. "N" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
percentage of participants
  Week 1 [N=75, 154] | 6.7 | 3.9
  Week 2 [N=71, 153] | 28.2 | 75.8
  Week 3 [N=70, 152] | 34.3 | 73.0
  Week 4 [N=170, 152] | 30.0 | 73.7
  Week 5 [N=68, 152] | 32.4 | 71.1
  Week 6 [N=66, 151] | 30.3 | 74.2
  Week 7 [N=66, 151] | 30.3 | 75.5
  Week 8 [N=65, 151] | 29.2 | 68.2
  Week 12 [N=62, 149] | 25.8 | 79.2
  Week 16 [N=61, 147] | 34.4 | 82.3
  Week 20 [N=58, 139] | 36.2 | 83.5
  Week 24 [N=58, 138] | 31.0 | 92.0
  Week 28 [N=57, 137] | 40.4 | 88.3
  Week 32 [N=55, 135] | 34.5 | 87.4
  Week 36 [N=54, 135] | 33.3 | 89.6
  Week 40 [N=52, 134] | 38.5 | 88.8
  Week 44 [N=51, 131] | 51.0 | 86.3
  Week 48 [N=48, 130] | 41.7 | 88.5
  Week 52 [N=38, 122] | 50.0 | 90.2

5. Secondary Outcome: Change in ITP-PAQ Physical Health Domain of Symptoms
Description: Change from Baseline in the Immune Thrombocytopenic Purpura (ITP) Patient Assessment Questionnaire (PAQ) physical health domain of symptoms. This domain has a range of 0 to 100, with higher scores indicating a better health-related quality of life.
  Model included fixed effects of baseline assessment, geographic region, treatment group, assessment week, splenectomy status and treatment group-by-assessment week interaction. Treatment group and splenectomy status are time-varying covariates.
Time Frame: Baseline and 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Units on a scale | 12.5 (2.1) | 16.0 (1.9)
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis — Significant level is set at 0.05

6. Secondary Outcome: Change in ITP-PAQ Physical Health Domain of Fatigue
Description: Change from Baseline in the Immune Thrombocytopenic Purpura (ITP) Patient Assessment Questionnaire (PAQ) physical health domain of fatigue. This domain has a range of 0 to 100, with higher scores indicating a better health-related quality of life. Model included fixed effects of baseline assessment, geographic region, treatment group, assessment week, splenectomy status and treatment group-by-assessment week interaction. Treatment group and splenectomy status are time-varying covariates.
Time Frame: Baseline and 52 weeks
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Units on a scale | 9.5 (3.2) | 11.2 (3.1)
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p = 0.3434, Mixed Models Analysis — Significant level is set at 0.05

7. Secondary Outcome: Change in ITP-PAQ Physical Health Domain of Bother
Description: Change from Baseline in the Immune Thrombocytopenic Purpura (ITP) Patient Assessment Questionnaire (PAQ) physical health domain of bother. This domain has a range of 0 to 100, with higher scores indicating a better health-related quality of life. Model included fixed effects of baseline assessment, geographic region, treatment group, assessment week, splenectomy status and treatment group-by-assessment week interaction. Treatment group and splenectomy status are time-varying covariates.
Time Frame: Baseline and 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Units on a scale | 13.0 (2.7) | 16.8 (2.5)
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis — Significant level is set at 0.05

8. Secondary Outcome: Change in ITP-PAQ Physical Health Domain of Activity
Description: Change from Baseline in the Immune Thrombocytopenic Purpura (ITP) Patient Assessment Questionnaire (PAQ) physical health domain of activity. This domain has a range of 0 to 100, with higher scores indicating a better health-related quality of life.
  Model included fixed effects of baseline assessment, geographic region, treatment group, assessment week, splenectomy status and treatment group-by-assessment week interaction. Treatment group and splenectomy status are time-varying covariates.
Time Frame: Baseline and 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Standard of Care | Romiplostim
Number analyzed (Participants) | 77 | 157
Units on a scale | 8.2 (3.7) | 17.1 (3.5)
Statistical Analysis 1: Comparison: Standard of Care vs Romiplostim; Test type: Superiority or Other; p = 0.0246, Mixed Models Analysis — Significant level is set at 0.05

ADVERSE EVENTS:
Time Frame: 52 week treatment period
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. 2 patients in Standard of Care (SOC) and 3 patients in the romiplostim arm did not receive the randomized treatment. 2 patients who were randomized to SOC and switched to romiplostim arm were counted in the Romiplostim arm.
Arm/Group | Standard of Care | AMG 531
Serious Adverse Events (participants affected / at risk) | 28/73 | 36/156
Other Adverse Events (participants affected / at risk) | 60/73 | 136/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=73) | AMG 531 (N=156)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 6
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatic fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
Sepsis (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Spinal haematoma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=73) | AMG 531 (N=156)
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Vertigo (Ear and labyrinth disorders) | 1 | 9
Abdominal pain (Gastrointestinal disorders) | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 6 | 16
Diarrhoea (Gastrointestinal disorders) | 4 | 21
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Gingival bleeding (Gastrointestinal disorders) | 5 | 9
Nausea (Gastrointestinal disorders) | 6 | 24
Vomiting (Gastrointestinal disorders) | 2 | 11
Chest pain (General disorders) | 4 | 6
Fatigue (General disorders) | 16 | 43
Influenza like illness (General disorders) | 0 | 8
Oedema peripheral (General disorders) | 3 | 15
Pain (General disorders) | 2 | 11
Pyrexia (General disorders) | 8 | 15
Hypersensitivity (Immune system disorders) | 4 | 3
Bronchitis (Infections and infestations) | 2 | 9
Gastroenteritis (Infections and infestations) | 1 | 10
Influenza (Infections and infestations) | 1 | 13
Nasopharyngitis (Infections and infestations) | 14 | 36
Sinusitis (Infections and infestations) | 1 | 13
Upper respiratory tract infection (Infections and infestations) | 6 | 18
Urinary tract infection (Infections and infestations) | 7 | 18
Contusion (Injury, poisoning and procedural complications) | 13 | 22
Procedural pain (Injury, poisoning and procedural complications) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 20
Dizziness (Nervous system disorders) | 6 | 21
Headache (Nervous system disorders) | 14 | 54
Paraesthesia (Nervous system disorders) | 0 | 9
Insomnia (Psychiatric disorders) | 9 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 19
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 10
Petechiae (Skin and subcutaneous tissue disorders) | 13 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 16
Rash (Skin and subcutaneous tissue disorders) | 5 | 13
Haematoma (Vascular disorders) | 9 | 12
Hypertension (Vascular disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.